CLINICAL TRIAL: NCT00955851
Title: A Study To Examine Serologic Response In Hospitalized Patients Receiving Polyvalent Pneumococcal Vaccine
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Juan Reyes, MD, George Washington University Medical Faculty Associates
Other Study IDs: 010902
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2009-08

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Lead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pneumonia patients: The study group will consist of individuals diagnosed with pneumonia and admitted to the Medicine ward under the Pneumonia Core Measure Protocol.
  Interventions: Other: Pre and post vaccination titers

INTERVENTIONS:
Other: Pre and post vaccination titers — Titers will be obtained pre vaccination and 4 weeks post vaccination

SUMMARY:
Investigators in the Division of Infectious Diseases and the Division of Hospital Medicine of The George Washington University Medical Center are carrying out a study to determine if hospitalized patients receiving the polyvalent pneumococcal vaccine during an acute illness develop an adequate antibody response. The study group will consist of individuals diagnosed with pneumonia and admitted to the Medicine ward under the Pneumonia Core Measure Protocol, which assigns appropriate patients for vaccination based on the current guidelines from the Advisory Committee on Immunization Practices (ACIP).

ELIGIBILITY:
Inclusion Criteria:

* Males or female patients ages 18 or older
* Diagnosis of pneumonia requiring hospitalization
* Admission to the Medicine Ward under the Pneumonia Core Measure protocol
* Eligible to receive standard of care pneumococcal vaccine by the treating physician
* Able to receive an injection
* Able to provide informed consent

Exclusion Criteria:

* Preexisting history of immunosuppression, to include any of the following: HIV/AIDS, Chronic corticosteroid use, Malignancy requiring myeloablative chemotherapy, Hematologic malignancy, History of solid organ or stem cell transplant
* Pregnancy
* Receipt of pneumococcal vaccine within the last 5 years
* Prior history of hypersensitivity reaction to the vaccine
* Unable to return for follow-up testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have been admitted to the Medicine Ward under the Pneumonia Core Measure Protocol as stated by the Joint Commission, and who receive the polyvalent pneumococcal vaccine as an inpatient as indicated by ACIP guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
A change in the pre- and post-vaccination pneumococcal serotype-specific IgG concentration from baseline will be considered protective based on the laboratory reference range. | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington University Hospital, Washington D.C., District of Columbia, United States